CLINICAL TRIAL: NCT00169819
Title: A Randomized Trial Comparing Same Day Discharge and a Single Bolus of Abciximab to Overnight Hospitalization and Bolus + Perfusion Abciximab After Uncomplicated Trans-Radial Coronary Artery Stenting
Brief Title: EArly Discharge After Transradial Stenting of CoronarY Arteries: The EASY Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H4S-CA-0050; ISRCTN72335887
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Artery Disease; Ischemia
Keywords: Same day discharge; Trans-radial; Coronary artery stenting; Abciximab bolus
MeSH Terms: conditions — Coronary Artery Disease; Ischemia | interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Abciximab

SUMMARY:
HYPOTHESES

* Discharge on the same day after uncomplicated trans-radial coronary artery stenting is safe and effective.
* Hospitalized patients can be safely returned to the referring center the same day following trans-radial coronary artery stenting.
* Abciximab given as a single bolus with optimal trans-radial coronary artery stenting is as safe and effective as bolus + 12 hrs perfusion and does not hamper early discharge.
* Same-day discharge is cost-effective and increases patient satisfaction.

OBJECTIVES AND END-POINTS

The objectives of the present study are to assess the effectiveness and safety of same day hospital discharge after uncomplicated coronary artery stenting when a single bolus of Abciximab is used. The primary end-point of the study is the composite of death, myocardial infarction, repeat hospitalization, urgent revascularization, severe thrombocytopenia, access site complications and major bleedings at 30 days following stent implantation.

The secondary end-point is the composite of death, myocardial infarction, repeat target vessel revascularization at 30 days, 6 months and 1 year following stent implantation. Other secondary end-points include the total hospital stay (days) between the index procedure and the first 30 days follow-up, the number of unsolicited medical visits in relation with the percutaneous procedure, index of patient satisfaction and direct and indirect costs.

DETAILED DESCRIPTION:
Despite significant improvements in clinical results associated with the current use of stenting and pharmacologic agents there has been little modification in hospitalization duration after percutaneous coronary interventions (PCI). The main reasons associated with prolonged hospitalization after PCI remain 1) the fear of abrupt vessel closure and its associated morbidity 2) the need for prolonged bed rest in case of femoral approach even after use of device closures.

The introduction of coronary stents has been associated with a dramatic decrease in vessel closure once it was recognized that stent deployment required higher pressure balloon inflation and increased antiplatelet therapy. Trans-radial coronary interventions appear safer and more cost-effective than femoral PCI. However, the current use of IIb-IIIa inhibitors prohibits the early discharge of patients following PCI because their pharmacology generally imposes to pursue drug infusion between 18 and 24 hrs following PCI which does not allow same day discharge from the hospital. With Abciximab, however, pharmacologic data indicate that prolonged platelet inhibition (≥ 80%) occurs after a single bolus. Based on the EPIC trial results, it has been recommended to prolong platelet inhibition by a 12 hrs perfusion. By analyzing carefully the EPIC trial results, we hypothesized that after optimal stenting result, a single bolus of Abciximab would suffice. We aim to demonstrate that (1) with trans-radial coronary stenting at least 50% of the entire population referred for PCI could be safely discharged after a few hours observation; (2) a single bolus of Abciximab is at least as effective as current recommended treatment with a bolus + 12 hrs perfusion after uncomplicated stenting. This new regimen could significantly affect current practice, decrease hospital costs and increase patient satisfaction after PCI.

STUDY DESIGN

A prospective randomized single-center study comparing same day hospital discharge to overnight hospitalization after uncomplicated trans-radial coronary artery stenting. Out-patients will be randomized after successful stent implantation to same day discharge or will remain hospitalized at Laval Hospital until the next morning. Hospitalized patients will be randomized after successful stent implantation to either same day discharge at home or to overnight hospitalization (either at the referring center or at Laval Hospital). All eligible patients will be treated with Abciximab that will be administered according to 2 different arms: For patients randomized to same-day discharge, only a bolus of Abciximab will be given, whereas for all remaining patients, Abciximab will be given according to current practice i.e. bolus + 12 hrs perfusion. All patients which will not be eligible post-PCI will enter a registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented ischemic coronary artery disease and scheduled for possible coronary artery stenting are eligible.
* Patient must be > 18 years of age.
* Patient and treating interventional cardiologist agree for randomization.
* Patient will be informed of the randomization process and will sign an informed consent.
* Diagnostic and therapeutic intervention performed through trans-radial/ulnar artery approach.

Exclusion Criteria:

CLINICAL:

* Patients with recent (< 72 hrs) Q-wave (ST elevation) acute myocardial infarction.
* History of LV ejection fraction ≤ 30%.
* Unstable clinical condition.
* Any complication compromising ambulation
* Concurrent participation in other investigational study requiring prolonged hospitalization
* Required prolonged hospitalization
* In-cath lab transient vessel closure
* Resuscitation per PCI
* Hemodynamic collapse during PCI
* Severe entry site complication upon investigator decision
* Social isolation
* Serious cognitive disorders
* Femoral sheath (artery)
* Persisting chest pain
* No ASA prior PCI
* Allergy to ASA or thienopyridines precluding treatment for 30 days
* Any significant blood dyscrasia
* PCI without stent implantation (except for bifurcation lesion or re-dilatation for in-stent restenosis)
* International Normalised Ratio (INR) > 2.0
* Contraindication to Reopro administration

ANGIOGRAPHIC

* Residual dissection of grade ≥ B of NHBLI classification.
* Compromised or sub-occluded branch with diameter ≥ 1 mm.
* Timi < 3 post-stenting
* Thrombus post-PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2003-10; Study Completion 2006-04

PRIMARY OUTCOMES:
Death, Q & non-Q myocardial infarction (MI), urgent revascularization, repeat hospitalization, severe thrombocytopenia, access site complications, major bleedings, at 30-days.

SECONDARY OUTCOMES:
Death, Q & non-Q MI, repeat target vessel revascularization at 30-days, 6 and 12 mo. Length of hospital stay & unsolicited medical visits at 30-days. Patient satisfaction within 24 hrs and at 30 days, 6 and 12 mo. Direct/indirect cost.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD, PhD, Principal Investigator — Laval Hospital Research Center
Locations (1):
- Laval Hospital Research Center, Sainte-Foy, Quebec, Canada

REFERENCES:
- [Result] Bertrand OF, De Larochelliere R, Rodes-Cabau J, Proulx G, Gleeton O, Nguyen CM, Dery JP, Barbeau G, Noel B, Larose E, Poirier P, Roy L; Early Discharge After Transradial Stenting of Coronary Arteries Study Investigators. A randomized study comparing same-day home discharge and abciximab bolus only to overnight hospitalization and abciximab bolus and infusion after transradial coronary stent implantation. Circulation. 2006 Dec 12;114(24):2636-43. doi: 10.1161/CIRCULATIONAHA.106.638627. Epub 2006 Dec 4. PMID 17145988
- [Derived] Rinfret S, Kennedy WA, Lachaine J, Lemay A, Rodes-Cabau J, Cohen DJ, Costerousse O, Bertrand OF. Economic impact of same-day home discharge after uncomplicated transradial percutaneous coronary intervention and bolus-only abciximab regimen. JACC Cardiovasc Interv. 2010 Oct;3(10):1011-9. doi: 10.1016/j.jcin.2010.07.011. PMID 20965458